CLINICAL TRIAL: NCT00006135
Title: Phase III Randomized Study of Oral Acyclovir in Infants With Herpes Simplex Virus Infection Limited to Skin, Eyes, and Mouth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Alabama at Birmingham (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/15334; UAB-CASG-104
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Herpes Simplex
Keywords: herpes simplex virus infection; herpesvirus infection; immunologic disorders and infectious disorders; rare disease; viral infection
MeSH Terms: conditions — Herpes Simplex; Herpesviridae Infections; Immune System Diseases; Communicable Diseases; Rare Diseases; Virus Diseases | interventions — Acyclovir

INTERVENTIONS:
Drug: acyclovir

SUMMARY:
OBJECTIVES:

I. Determine the efficacy of long term suppressive therapy with oral acyclovir in infants with herpes simplex virus infection limited to skin, eyes, and mouth.

II. Determine the neurologic outcome in these patients when treated with this regimen.

III. Evaluate the significance of a positive cerebrospinal fluid (CSF) polymerase chain reaction (PCR) result when all other CSF parameters remain normal in these patients.

IV. Correlate the time to first positive CSF PCR result in the first 12 months of life with clinical neurological assessment in these patients when treated with this regimen.

V. Determine whether the continuous administration of this drug suppresses recurrent skin lesions in these patients.

VI. Determine the safety of this regimen in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, double blind, placebo controlled, multicenter study.

All patients undergo a lumbar puncture and then receive acyclovir IV every 8 hours on Days 1-14. On Day 12, patients may undergo a lumbar puncture (at discretion of investigator). Whole blood is obtained for herpes simplex virus PCR analysis. Upon completion of intravenous therapy, patients with a negative CSF PCR are randomized to one of two treatment arms.

Arm I: Patients receive oral acyclovir three times daily for 6 months.

Arm II: Patients receive placebo three times daily for 6 months.

In case of cutaneous recurrence during the first 12 months of the study, patients receive open label oral acyclovir (if CSF PCR is negative) or acyclovir IV (if CSF PCR is positive) for 5 days. Patients may or may not continue on study drug following this treatment.

Patients are followed at 6, 12, 24, 36, 48, and 60 months of age.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Infants diagnosed with herpes simplex virus infection limited to skin, eyes, and mouth; HSV-1 or HSV-2 isolated from cutaneous lesions, conjunctivae, or oropharynx (presence of skin lesions not required); normal CSF indices: WBC less than 22/mm3 and protein less than 115 mg/dL for term infants OR WBC less than 25/mm3 and protein less than 220 mg/dL for preterm infants; no evidence of CNS involvement by CT with contrast, MRI with gadolinium, or head ultrasound; no visceral dissemination (normal liver function tests, normal chest x-ray, etc.); negative CSF PCR result

Birth weight at least 800 grams

--Prior/Concurrent Therapy--

No concurrent nursing from a mother who is receiving acyclovir, valacyclovir, or famciclovir for longer than 120 hours or 5 days; no prior prophylactic acyclovir for risk of herpes simplex virus infection

--Patient Characteristics--

Renal: Creatinine no greater than 1.5 mg/dL

Cardiovascular: No prior grade 3 or 4 intraventricular hemorrhage

Other: No infants known to be born to HIV-positive women

Ages: 0 Years to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66
Dates: Start 1997-06

CONTACTS AND LOCATIONS:
Overall Officials: David W. Kimberlin, Study Chair — University of Alabama at Birmingham
Locations (27):
- United States (25):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of Arkansas, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital and Health Center, San Diego, California
  - Stanford University, Stanford, California
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Tulane University Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis Children's Hospital, St Louis, Missouri
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Children's Hospital, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Medical Center at Knoxville, Knoxville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical School, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba-Winnipeg, Winnipeg, Manitoba